CLINICAL TRIAL: NCT00548145
Title: The Clinical Study of Pitavastatin Treatment for Group of Mild to Moderate Alzheimer's Disease
Acronym: PIT-ROAD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Osaka University (Other)
Collaborators: Kowa Company, Ltd. (Industry)
Responsible Party: Principal Investigator, Hiroaki Kazui, M.D.Ph.D, Osaka University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OSK-07098
Record Dates: First submitted 2007-10-22; First posted 2007-10-23 (Estimated); Results first posted 2012-06-14 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-05

CONDITIONS: Alzheimer Disease; Hypercholesterolemia
Keywords: Pitavastatin; Statins; Donepezil; Alzheimer's Disease; Hypercholesterolemia; ADAS-Jcog; Alzheimer Disease (MMSE 15-23 and CDR1 or 2)
MeSH Terms: conditions — Alzheimer Disease; Hypercholesterolemia | interventions — pitavastatin; colestimide

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Pitavastatin
- 2 (Active Comparator)
  Interventions: Drug: cholesterol-lowering medicine other than statin(e.g.,Ezetimibe,Colestimide)

INTERVENTIONS:
Drug: Pitavastatin — 2 mg by orally/day Duration: 12 months
  Arms: 1
Drug: cholesterol-lowering medicine other than statin(e.g.,Ezetimibe,Colestimide) — duration: 12 months
  Arms: 2

SUMMARY:
Some studies suggest that statin medications may be effective against Alzheimer's disease. However, this has not been proven. The purpose of this study is to evaluate the efficacy of pitavastatin in patients with mild to moderate Alzheimer's disease and hypercholesterolemia.

DETAILED DESCRIPTION:
The PIT-ROAD study will include 50 patients who have taken donepezil more than 3 months stably. This study will see how the use of a particular statin medication, pitavastatin, affects ADAS-Jcog score etc. and cholesterol.

Participants will be given a full information of the study and written informed consent should be obtained before entering the study. Participants will take part in 5 visits over the course of 12 months. If participants have taken cholesterol lowering drug, they will have wash-out period at least 4weeks. Participants will undergo 8 tests (ADAS-Jcog etc., baseline and month 12 visits), complete a medical history questionnaire (baseline), complete medication side effect review through questionnaire and/or blood sample (all visits). Participants will be randomly assigned to receive either pitavastatin or other cholesterol lowering medication for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Alzheimer's Disease patients (15 ≤ MMSE total score ≤ 23, CDR "1" or "2")
* Patients with hypercholesterolemia
* Patients who have taken donepezil more than 3 months stably
* Both patients and care-givers must be more than 20 years old

Exclusion Criteria:

* Women with pregnancy or breast-feeding
* Malignant tumor
* Cerebrovascular disorder or myocardial infarction prior to 12 weeks
* Heart failure [New York Heart Association (NYHA) class III or IV]
* Hepatic or renal dysfunction
* Severe hypertension
* Hypothyroidism, hereditary muscular disease, history of drug-induced myopathy
* Current involvement in another investigational drug study
* Alcoholism, drug abuse

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2007-11; Primary Completion 2011-10 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hiroaki Kazui, Ph.D., Principal Investigator — Osaka University Hospital
Locations (1):
- Osaka University Hospital, Suita, Osaka, Japan

REFERENCES:
- See also: Related Info — http://www.med.osaka-u.ac.jp/pub/psy/www/en/index.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Hyperlipidemia patients with mild to moderate Alzheimer's disease(MMSE15～23)
Groups:
- Cholesterol-lowering Medicine Other Than Statin: duration: 12 months
Period: Overall Study
Arm/Group | Pitavastatin | Cholesterol-lowering Medicine Other Than Statin
Started | 18 | 20
Completed | 17 | 16
Not Completed | 1 | 4
Not completed — Death | 0 | 1
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Physician Decision | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pitavastatin | Cholesterol-lowering Medicine Other Than Statin | Total
Number analyzed (Participants) | 18 | 20 | 38
Age Continuous [Mean (Standard Deviation); unit: years] | 75.8 (7.2) | 75.3 (7.7) | 75.5 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 18 | 35
  Male | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Alzheimer's Disease Assessment Scale-cognitive Component-Japanese Version(ADAS-Jcog)
Description: Alzheimer's Disease Assessment Scale-cognitive component-Japanese version is a cognitive test for Alzheimer's disease. This test includes some aspects that assess memory ,orientation, language, praxis, and so on. The possible range of this test is 0-70 points.Higher total points indicate more impairment.
Time Frame: baseline and 12 months
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Pitavastatin | Cholesterol-lowering Medicine Other Than Statin
Number analyzed (Participants) | 17 | 16
scores on a scale
  baseline | 18.59 (6.13) | 19.50 (5.61)
  12month | 20.20 (9.31) | 20.59 (7.91)

2. Secondary Outcome: MMSE, Neuropsychiatric Inventory, GDS-15, Zarit Burden Scale, Physical Self-Maintenance Scale, IADL, Everyday Memory Checklist, TC, HDL-C, Non HDL-C*, Apo A1, Apo B, Apo E *: Non HDL-C = (TC) - (HDL-C)
Description: Mini-Mental State Examination(MMSE),Geriatric Depression Scale-15(GDS-15),Instrumental Activities of Daily Living Scale(IADL),Total Cholesterol(TC)
Time Frame: baseline and 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Pitavastatin | Cholesterol-lowering Medicine Other Than Statin
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/20
Other Adverse Events (participants affected / at risk) | 0/18 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other